CLINICAL TRIAL: NCT05230225
Title: Electronic Physician Notification to Facilitate the Recognition and Management of Severe Aortic Stenosis: The DETECT AS Trial
Acronym: DETECT AS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, Sammy Elmariah, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022P000016
Record Dates: First submitted 2022-01-13; First posted 2022-02-08 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Aortic Stenosis
Keywords: Aortic Valve Stenosis; Aortic Valve Disease; Heart Valve Diseases; Heart Diseases; Cardiovascular Diseases; Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Disease; Heart Valve Diseases; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Notification Letter Arm (Experimental): Providers that will receive an electronic Physician Notification Letter.
  Interventions: Behavioral: Physician Notification Letter
- Control Group (No Intervention): Providers that will not be contacted.

INTERVENTIONS:
Behavioral: Physician Notification Letter — Receiving the electronic Physician Notification Letter to highlight echocardiography results that are consistent with or may be consistent with severe AS and to be reminded of ACC/AHA Clinical Practice Guideline recommendations regarding the management of severe AS.
  Arms: Notification Letter Arm

SUMMARY:
The DETECT AS Trial is a randomized clinical trial and quality improvement initiative that seeks to investigate the impact of electronic provider notification of severe aortic stenosis (AS) on its management, on the utilization of aortic valve replacement (AVR), and on ethnic and racial disparities in AVR utilization.

After the investigators identify patients in whom echocardiography shows severe aortic stenosis, defined by an aortic valve area (AVA) <1.0cm2, the ordering provider of the echocardiogram will then be randomly assigned to either the intervention group or to the control group. Providers randomly assigned to the intervention group will be sent an electronic (email or message via the electronic health record) physician notification for every one of their patients with severe aortic stenosis on TTE. Electronic notification will also highlight relevant ACC/AHA Clinical Practice Guideline recommendations regarding the management of severe AS. No intervention will be performed for patients belonging to physicians assigned to the control group.

The primary endpoint will be AVR utilization, defined as the proportion of patients with a clinical indication for severe AS that undergo AVR. Clinical indications will be based upon the 2020 AHA/ACC Clinical Practice Guidelines for Valvular Heart Disease.

Secondary end-points will be mortality, heart failure hospitalization, TTE utilization/surveillance, AS billing code diagnosis, and cardiology/Heart Valve Team referral. Pre-defined subgroup analyses will be performed to assess AVR utilization among women, racial/ethnic minority groups, low-gradient AS, cardiologist and non-cardiologist ordering provider, and inpatient and outpatient practice settings.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with severe aortic stenosis having an aortic valve area of less than or equal to 1.0cm2.

Exclusion Criteria:

* Subjects with bioprosthetic or mechanical valves in the aortic position

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 940 (Estimated)
Dates: Start 2022-02-09 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Establish impact of electronic physician notification letter on the likelihood of AVR utilization for patients with a clinical indication for severe AS | 1 year
  Determining whether an electronic physician notification letter improves recognition and management of severe AS through its impact on the utilization of aortic valve replacement, which is defined as the proportion of patients with a clinical indication for severe AS that undergo AVR. We will utilize electronic notification letter to highlight TTE results that are consistent with or may be consistent with severe AS and providers will also be reminded of ACC/AHA Clinical Practice Guideline recommendations regarding the management of severe AS.

SECONDARY OUTCOMES:
Impact on mortality rate | 1 year
  Establishing the mortality rate among patients with severe AS followed until one year after symptom onset. Using data analysis we will investigate the impact of physician notification letters on recognition and management of AS based on it's effect on mortality rate.
Impact on rate of heart failure hospitalization | 1 year
  Determining the rate of heart failure hospitalizations among patients with severe AS followed until one year after symptom onset. Using data analysis we will investigate the impact of physician notification letters on recognition and management of AS based on it's effect on likelihood of heart failure hospitalization.
Impact on rate of trans-thoracic echocardiogram utilization and frequency of surveillance | 1 year
  Identifying all trans-thoracic echocardiograms ordered by physicians for patients with severe AS until one year after symptom onset in order to Investigate the impact of physician notification letters on the number of follow up echocardiograms ordered and the frequency of surveillance.
Impact on proportion of patients referred to Cardiology/Heart Valve Team | 1 year
  Determining when patients with severe AS get referred to a Cardiology/Heart valve team. Providers receive physician notification letters detailing ACC/AHA Clinical Practice Guideline Recommendations that suggest patients with severe valvular heart disease should be evaluated by a Multidisciplinary Heart Valve Team when intervention is considered. Using data analysis we will investigate the impact of physician notification letters on rate of referral and time to referral to a Cardiology/Heart Valve Team.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tanguturi VK, Abou-Karam R, Cheng F, Duan R, Inglessis-Azuaje I, Langer NB, Yucel EN, Passeri JJ, Hung JW, Elmariah S. Electronic Provider Notification to Facilitate the Recognition and Management of Severe Aortic Stenosis: A Randomized Clinical Trial. Circulation. 2025 May 27;151(21):1498-1507. doi: 10.1161/CIRCULATIONAHA.125.074470. Epub 2025 Mar 30. PMID 40159132
- [Derived] Abou-Karam R, Tanguturi V, Cheng F, Elmariah S. Electronic physician notification to facilitate the recognition and management of severe aortic stenosis: Rationale, design, and methods of the randomized controlled DETECT AS trial. Am Heart J. 2024 Oct;276:39-48. doi: 10.1016/j.ahj.2024.06.009. Epub 2024 Jun 29. PMID 38950668